CLINICAL TRIAL: NCT04958187
Title: An Open Label, Single-Dose Study to Evaluate the Safety and Pharmacokinetics of ANG-3777 Injected Intravenously in Stable Adult Maintenance Hemodialysis Subjects
Brief Title: Study to Evaluate the Pharmacokinetics of ANG-3777 in Hemodialysis Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Angion Biomedica Corp (Industry)
Collaborators: Nucleus Network Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANG3777-HD-103
Record Dates: First submitted 2021-06-30; First posted 2021-07-12 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Hemodialysis
MeSH Terms: interventions — terevalefim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ANG-3777 (Experimental): Administered IV as a single dose over 30 minutes on Day 1, greater than 24 hours before receiving scheduled hemodialysis (HD).
  Interventions: Drug: ANG-3777

INTERVENTIONS:
Drug: ANG-3777 — Arm assigned to this intervention will receive 2 mg/kg, IV
  Other Names: Hepatocyte growth factor mimetic

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of a single-dose of ANG-3777 in subjects with renal failure receiving maintenance hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female subjects, 18 to 75 years of age at time of informed consent who have been on maintenance HD 3 times a week for at least 3 months prior to signing informed consent.
2. Must receive HD 3 times a week.
3. Target post-dialysis body weight < 125 kg.
4. Have laboratory parameters at Screening as follows:

   1. Serum albumin ≥ 3.0 g/dL
   2. Blood hemoglobin ≥ 9.0 g/dL
   3. Serum liver transaminases (alanine aminotransferase [ALT], aspartate aminotransferase [AST]) < 2× the upper limit of normal
5. Have adequate single pool urea (Kt/V ≥ 1.2) for the 2 consecutive readings in the months preceding the Screening Visit.
6. Subjects will not be allowed to start any new medications during the study period (i.e., from treatment assignment to the follow-up visit) except in case of a medical emergency (the subject may be removed from the study accordingly as decided by the Principal Investigator [PI] and sponsor).
7. Subjects should be on stable doses of medications for at least 2 weeks preceding check-in to the research unit except medications used to manage co-morbidities associated with dialysis, e.g., Epogen, vitamin D analogs, and Venofer.
8. Women of childbearing potential will not be breast feeding and must have a negative serum pregnancy test at Screening and Day -1.
9. Women of childbearing potential must use 2 forms of effective birth control (at least one barrier method) during the study and for 31 days after end of infusion. Men will be required to use condoms for the duration of study and for 7 days after study discharge.
10. In the opinion of the investigator, the subject is capable of understanding and complying with the protocol. Subjects must have signed and dated the ICF prior to performance of any study related procedure including Screening procedures.
11. Must be receiving HD via an arterio-venous fistula or an arterio-venous graft with no access procedure performed within 1 month prior to receiving study drug.

Exclusion Criteria:

1. Subjects treated with the cytochrome P450 1A2 (CYP1A2) inhibitors ciprofloxacin (Cipro®) or fluvoxamine (Luvox®) within 14 days prior to anticipated first dose of study medication.
2. Ongoing infections or the use of anti-infective medications within 2 weeks prior to Screening.
3. History of previous organ transplant or known liver disease.
4. Have ongoing drug abuse/dependence (including alcohol) or recent history (within the past 5 years) of, or treatment for, alcohol or drug abuse.
5. Positive serum test for alcohol at Screening or on Day -1.
6. Positive drugs of abuse test at Screening (serum) or on Day -1 (saliva).
7. Current smokers who smoke > 5 cigarettes a day (serum cotinine levels ≥ 10 ng/mL) are excluded. Note: Cotinine is tested at Screening only. Every effort should be made to recruit nonsmokers; at least 8 subjects in this study should be nonsmokers.
8. Subjects with an active malignancy, suspicion of active malignancy by history or physical examination, or history of solid, metastatic, or hematologic malignancy with the exception of basal or squamous cell carcinoma of the skin that has been removed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Measure the pharmacokinetic (PK) parameters of a single dose of ANG-3777 including, but not limited to: Tmax | Day 1 and Day 2
Measure the pharmacokinetic (PK) parameters of a single dose of ANG-3777 including, but not limited to: Cmax | Day 1 and Day 2
Measure the pharmacokinetic (PK) parameters of a single dose of ANG-3777 including, but not limited to: AUC(0-last) and AUC(0-inf) | Day 1 and Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K. Ries, MD, Principal Investigator — Nucleus Network Ltd
Locations (1):
- Hennepin County Medical Center (HCMC), Minneapolis, Minnesota, United States